CLINICAL TRIAL: NCT05936866
Title: Effect of Antenatal Pelvic Floor Stretching Vs Strengthening Exercises on Maternal Birth Outcomes in Primigravida
Brief Title: Effects of Antenatal Exercises on Maternal Birth Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/01537 Omama Sadaf
Record Dates: First submitted 2023-06-26; First posted 2023-07-10 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Pregnancy Related
Keywords: Pregnancy Related; Pelvic Floor Muscle Weakness; Delivery Delayed

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pelvic floor stretching (Experimental): Pelvic floor stretching exercises
  Interventions: Other: Pelvic floor stretching
- Pelvic floor strengthening (Active Comparator): Pelvic floor strengthening Exercises
  Interventions: Other: Pelvic floor strengthening

INTERVENTIONS:
Other: Pelvic floor stretching — Week 1 to 4: Pelvic floor muscles awareness, Breathing exercises , seated pelvic tilts, cat stretches, seated hip openers (2 sets, 8 reps, sustained for 6 seconds) Week 5 to 8: Pelvic floor muscles awareness, Breathing exercises ,seated pelvic tilts, cat stretches, Seated hip openers, Relaxed Frog (2 sets, 8 reps, sustained for 6 seconds) Week 9 to 13: Pelvic floor muscles awareness, Breathing exercises, seated pelvic tilts, cat stretches, Seated hip openers, Relaxed Frog side lying clamshells, mini squats with support (2 sets, 9 reps, sustained for 7 seconds)
  Arms: Pelvic floor stretching
Other: Pelvic floor strengthening — Week 1 to 4: Pelvic floor muscles awareness, Breathing exercises, 2 Sets of 10 Reps for pelvic floor squeeze and release Seated marching with elastic band with pelvic floor squeeze.
  Week 5 to 8: 2 sets x 9 Reps for Pelvic floor squeeze and release, Seated marching with elastic band with pelvic. 2 Sets x 8 Reps for bridging with pelvic floor squeeze, side lying hip circles Week 9 to 13: 2 sets 10 reps for Pelvic floor squeeze-and-release, Seated marching with elastic band with pelvic floor squeeze, pelvic bridging with pelvic floor squeeze, side lying hip circles with pelvic floor squeeze. 2 sets, 8 reps for . side lying Clamshells with resistance band and pelvic floor squeeze and plie squats with pelvic floor squeeze
  Arms: Pelvic floor strengthening

SUMMARY:
The study is aimed to determine the effects of pelvic floor stretching Vs strengthening on maternal birth outcomes and postpartum urogenital distress in primigravida.

DETAILED DESCRIPTION:
The effects of pelvic floor muscle exercises on the symptoms of postpartum urinary distress is not known, so there is a need to determine whether strengthening or stretching of pelvic floor muscles help in reducing the risk of developing urogenital distress in postpartum period of females. The positive effect of pelvic floor muscle training on duration of labor and maternal birth outcomes is understood. As stated in a systemic review of pelvic floor interventions during pregnancy. The researches done on effect of pelvic floor muscle exercises, included once a week supervised session of sustained pelvic floor muscle contractions with rest intervals and fast contractions with respective rest intervals along with daily home sessions of the same exercises.

ELIGIBILITY:
Inclusion Criteria:

* Primigravida

Exclusion Criteria:

* Any Contraindications to performing an exercise during pregnancy based on recommendations of the American College of Obstetricians and Gynecologists (ACOG)
* females opting for Elective C section

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 42 (Actual)
Dates: Start 2023-06-13 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2023-12-21 (Actual)

PRIMARY OUTCOMES:
Mode of delivery | 13th Week
  Changes from the baseline outcome of Mode of Delivery will be taken from the delivery and labor records of the patients and also from the consultant Gynecologist.
Duration of labour | 13th Week
  Changes from the baseline outcome of Duration of labour will be taken from the delivery and labor records of the patients and also from the consultant Gynecologist. It will be measured in minutes/hours.
Number of vaginal inductions | 13th Week
  Changes from the baseline outcome of Number of vaginal inductions will be taken from the delivery and labor records of the patients and also from the consultant Gynecologist. It will be measured in minutes/hours.

SECONDARY OUTCOMES:
Urogenital Distress Inventory | 15th Week
  UDI-6 is a widely used tool for the assessment of quality of life and symptoms of urinary incontinence in women. It is the short form which consists of 6 questions which are: frequent urination, leakage related to feeling of urgency, leakage related to activity, coughing or sneezing. Amount of drops of leakage, difficulty emptying the bladder and pain and discomfort in the lower abdominal or genital area. Scoring: Item responses are assigned values of 0 for "not at all," 1 for "slightly," 2 for "moderately," and 3 for "greatly." The average score of items responded to is calculated. The average, which ranges from 0 to 3, is multiplied by 33 1/3 to put scores on a scale of 0 to 100.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Ehsan, PP-DPT, Principal Investigator — Riphah International University
Locations (1):
- Doctors hospital, Abbottabad, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No